CLINICAL TRIAL: NCT02592525
Title: Implementing Shared Decision Making in Interprofessional Home Care Teams : a Stepped Wedge Cluster Randomized Trial
Brief Title: Implementing Shared Decision Making in Interprofessional Home Care Teams
Acronym: IPSDM-SW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, France Legare, Canada Research Chair in Implementation of Shared Decision Making in Primary Care, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015-2016 01-01-E
Record Dates: First submitted 2015-10-28; First posted 2015-10-30 (Estimated); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Aging
MeSH Terms: interventions — Health Personnel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cluster A (Experimental): IP-SDM training for health professionals (intervention at 4 months)
  Interventions: Behavioral: IP-SDM training for health professionals
- Cluster B (Experimental): IP-SDM training for health professionals (intervention at 11 months)
  Interventions: Behavioral: IP-SDM training for health professionals
- Cluster C (Experimental): IP-SDM training for health professionals (intervention at 18 months)
  Interventions: Behavioral: IP-SDM training for health professionals
- Cluster D (Experimental): IP-SDM training for health professionals (intervention at 25 months)
  Interventions: Behavioral: IP-SDM training for health professionals

INTERVENTIONS:
Behavioral: IP-SDM training for health professionals — Multifaceted SDM training program for providers: i) 1.5-hour online tutorial, ii) 3.5-hour skills building workshop; iii) video-clip demonstrating SDM in the context of an IP home care team with an aging adult making a decision about location of care (to be used with clients and providers as well); and iv) performance feedback to providers (role play during the workshop).

SUMMARY:
This study will train health providers in home care teams across Quebec in shared decision making about the decision to stay at home or move to another location. This decision is one of the toughest for older Canadians. Decisions that are informed, shared and supported produce better results. An interprofessional approach to shared decision making is when older persons and their caregivers are supported by not just one but by all the professionals involved in their care.The impact of the training program in interprofessional shared decision making (IPSDM) above that of the passive dissemination of a decision guide will be assessed by measuring to what extent older persons caregivers say they took active part in the decision-making process.

Other outcome measures will be:

i) what option they chose, whether they feel conflict or regret about their decision, and the burden of care they feel; ii) the quality of life of clients;

ELIGIBILITY:
Inclusion Criteria:

Clients or caregivers of clients :

* Aged ≥65 years;
* Receiving care from the IP home care team of the enrolled CISSS/CIUSSS
* Have made a decision about whether to stay at home or move to another location during the recruitment periods
* Are able to read, understand and write French or English
* Can give informed consent

In the case clients are not able to provide informed consent, their caregiver will be eligible.

Exclusion Criteria:

* Clients who are not able to provide informed consent and who don't have a caregiver

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 653 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Assumed Role in decision making | 7 months
  To assess the proportion of caregivers reporting an active role, a modified version of the Control Preferences Scale designed to assess the role assumed in the decision making process will be used. The scale consists of a single question and is the one most frequently used in studies assessing the implementation of SDM in clinical practice.

SECONDARY OUTCOMES:
Patient involvement in decision making | 7 months
  Assessed with the Dyadic-OPTION scale, a 12-item self-administered instrument that assesses 12 specific SDM behaviours during the decision-making process
Decisional Regret | 7 months
  Assessed with the Decisional Regret Scale
Decisional Conflict | 7 months
  Assessed with the Decisional Conflict Scale
Health-related quality of life | 7 months
  Assessed with two subscales (Social isolation and Emotional reactions) of the HR-QoL questionnaire from the Nottingham Health Profile, clients only
Burden of care | 7 months
  Assessed with the Zarit Burden Inventory Scale (ZBI), caregivers only
Preferred and chosen option (remain at home or move to another location) | 7 months
  Questionnaire assessing the prefered and chosen option

CONTACTS AND LOCATIONS:
Overall Officials: France Légaré, Ph. D., Principal Investigator — Laval University
Locations (1):
- Centre de recherche sur les soins et les services de première ligne de l'Université Laval (CERSSPL-UL), Québec, Quebec, Canada

REFERENCES:
- [Derived] Adisso EL, Taljaard M, Stacey D, Briere N, Zomahoun HTV, Durand PJ, Rivest LP, Legare F. Shared Decision-Making Training for Home Care Teams to Engage Frail Older Adults and Caregivers in Housing Decisions: Stepped-Wedge Cluster Randomized Trial. JMIR Aging. 2022 Sep 20;5(3):e39386. doi: 10.2196/39386. PMID 35759791
- [Derived] Legare F, Briere N, Stacey D, Lacroix G, Desroches S, Dumont S, Fraser KD, Rivest LP, Durand PJ, Turcotte S, Taljaard M, Bourassa H, Roy L, Painchaud Guerard G. Implementing shared decision-making in interprofessional home care teams (the IPSDM-SW study): protocol for a stepped wedge cluster randomised trial. BMJ Open. 2016 Nov 24;6(11):e014023. doi: 10.1136/bmjopen-2016-014023. PMID 27884857
- See also: Related Info — http://www.decision.chaire.fmed.ulaval.ca/